CLINICAL TRIAL: NCT01589627
Title: Contracture Reduction Following Distal Radius Fracture
Brief Title: Wrist Extension Dynasplint (WED) Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009.003
Record Dates: First submitted 2012-04-27; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Distal Radius Fracture; Wrist Contracture
Keywords: distal radius fracture; wrist contracture; dynasplint
MeSH Terms: conditions — Wrist Fractures

ARMS (2):
- experimental (Experimental): Patients will be treated with the Standard of Care physical therapy, NSAIDs as well as a Wrist Extension Dynasplint
  Interventions: Device: Wrist Extension Dynasplint
- Control (No Intervention): Patients will receive standard of care physical therapy and NSAIDS

INTERVENTIONS:
Device: Wrist Extension Dynasplint — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. The Knee Extension Dynasplint for the Experimental group will have tension chambers delivering therapeutic treatment from the device.
  Arms: experimental

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a dynamic splinting system for wrist extension contracture following a distal radius fracture.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture treated with surgical management and wrist flexion contracture upon follow up

Exclusion Criteria:

* Carpal Fractures (Scaphoid, Lunate, Hamate, and Trapezium)
* Radial nerve entrapment
* Arthrodesis
* Traumatic dislocation of the distal ulna

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximal active range of motion in wrist extension | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Berner, MD, Principal Investigator — Advanced Centers for Orthopaedic Surgery and Sports Medicine